CLINICAL TRIAL: NCT01448824
Title: A Phase 1 Study to Evaluate the Safety and Tolerability of LY2484595 SDSD-PG Tablets and the Effect of CYP3A Inhibition by Ketoconazole on the Pharmacokinetics of LY2484595 in Healthy Subjects
Brief Title: A Study of LY2484595 on Pharmacokinetics in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 14460; I1V-MC-EIAL (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-10-06; First posted 2011-10-07 (Estimated); Results first posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Healthy Participants
Keywords: Low High-density Lipoprotein (HDL); Cholesterol (HDL-C)
MeSH Terms: interventions — evacetrapib; Ketoconazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Part 1 (Cohort A): 100 mg, 1800 mg LY2484595, Placebo (Experimental): Period 1: Participants will receive either 100 milligrams (mg) LY2484595 tablets or placebo tablets once daily (QD) by mouth on Days 1 through 14 of Period 1.
  Washout period lasting ≥14 days.
  Period 2: Participants will receive either 1800 mg LY2484595 tablets or placebo tablets QD by mouth on Days 1 through 14 of Period 2.
  Interventions: Drug: LY2484595; Drug: Placebo
- Part 1 (Cohort B): 300 mg LY2484595, Placebo (Experimental): Participants will receive either 300 milligrams (mg) LY2484595 tablets or placebo tablets once daily (QD) by mouth on Days 1 through 14.
  Interventions: Drug: LY2484595; Drug: Placebo
- Part 1 (Cohort C): 600 mg LY2484595, Placebo (Experimental): Participants will receive either 600 milligrams (mg) LY2484595 tablets or placebo tablets once daily (QD) by mouth on Days 1 through 14.
  Interventions: Drug: LY2484595; Drug: Placebo
- Part 1 (Cohort D): 1200 mg LY2484595, Placebo (Experimental): Participants will receive either 1200 milligrams (mg) LY2484595 tablets or placebo tablets once daily (QD) by mouth on Days 1 through 14.
  Interventions: Drug: LY2484595; Drug: Placebo
- Part 2 (Cohort E): 100 mg LY2484595 ± 400 mg Ketoconazole (Experimental): Period 1: Participants will receive 100 milligrams (mg) LY2484595 tablet by mouth on Day 1 of Period 1.
  Washout period lasting ≥14 days.
  Period 2: Participants will receive 400 mg ketoconazole tablets once daily (QD) by mouth on Days 1 through 14 of Period 2. Participants will receive 100 mg LY2484595 tablet by mouth on Day 5 of Period 2.
  Interventions: Drug: LY2484595; Drug: Ketoconazole

INTERVENTIONS:
Drug: LY2484595 — Administered orally
Drug: Placebo — Administered orally
  Arms: Part 1 (Cohort A): 100 mg, 1800 mg LY2484595, Placebo; Part 1 (Cohort B): 300 mg LY2484595, Placebo; Part 1 (Cohort C): 600 mg LY2484595, Placebo; Part 1 (Cohort D): 1200 mg LY2484595, Placebo
Drug: Ketoconazole — Administered orally
  Arms: Part 2 (Cohort E): 100 mg LY2484595 ± 400 mg Ketoconazole

SUMMARY:
This is a 2-part study. Part 1 is to determine the safety and tolerability in healthy participants of increasing daily doses of LY2484595 for 14 days to achieve a blood level of LY2484595 much higher than what is needed for therapy. The amount of study drug that reaches the bloodstream and the time it takes for the body to get rid of it will be determined. The effect of the study drug on factors in the blood related to cholesterol will be measured.

Part 2 is to determine how ketoconazole affects how much of the study drug, LY2484595, gets into the bloodstream and how long it takes to get rid of it. Information about any side effects that may occur will also be collected.

DETAILED DESCRIPTION:
This study is a 2-part, multiple ascending dose (MAD) and drug drug interaction (DDI) study to evaluate the safety and tolerability and the effect of cytochrome P450 (CYP) 3A inhibition by ketoconazole on the pharmacokinetics of LY2484595 in healthy participants.

In the MAD portion (Part 1) of this study, participants in 4 cohorts (Cohorts A through D) will be randomized to receive either LY2484595 (5 ascending dose levels [100 to 1800 mg]) or placebo. Cohorts will have staggered starts ≥7 days from the previous cohort to allow for review of safety and tolerability. The total duration of Part 1 is approximately 13 weeks including screening.

Participants in Cohort A will participate in 2 periods separated by a washout period lasting ≥14 days. During Period 1, participants will receive the starting dose of LY2484595 (100 mg) or placebo once daily (QD) for 14 consecutive days. During Period 2, participants will receive the highest dose of LY2484595 (1800 mg) or placebo QD for 14 consecutive days. Participants will complete a follow-up visit ≥14 days after the last dose of study drug.

Participants in Cohorts B, C, and D will receive LY2484595 (300, 600, and 1200 mg LY2484595, respectively) or placebo QD for 14 consecutive days followed by a follow-up visit ≥14 days after last dose of study drug.

The DDI portion of this study (Part 2) will be open label and consist of 2 periods. The total duration of Part 2 is approximately 10 weeks. LY2484595 (100 mg) will be administered on Day 1 of Period 1 and on Day 5 of Period 2. In Period 2, ketoconazole (400 mg) will be administered QD for 14 consecutive days (13 days alone [Days 1 through 4 and 6 through 14] + 1 day with LY2484595 [Day 5]). There will be a ≥14-day washout period between dosing during Period 1 and Period 2. Participants will return for a follow-up visit ≥14 days after last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females, as determined by medical history and physical examination
* Female participants and women not of childbearing potential due to surgical sterilization (hysterectomy, bilateral oophorectomy, or tubal ligation) or menopause. Postmenopausal is defined as women age >45 with an intact uterus who have not taken hormones or oral contraceptives within the last year, and who have had either cessation of menses greater than or equal to 1 year or 6 to 12 months of spontaneous amenorrhea with follicle-stimulating hormone (FSH) >40 milli-international units per milliliter (40 international units per liter [IU/L]).
* Have a body mass index (BMI) between 18 to 32 kilograms per square meter (kg/m^2), inclusive
* Have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Have venous access sufficient to allow for blood sampling
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Have given written informed consent approved by Lilly and the institutional review board (IRB) governing the site

Exclusion Criteria:

* Are currently enrolled in, have completed or discontinued within the last 30 days from a clinical trial involving an investigational product, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have known allergies to LY2484595 or related compounds, contraindications to ketoconazole or related compounds, or allergies to any components of the formulations
* Are persons who have previously completed or withdrawn from this study or any other study investigating LY2484595 and have previously received the investigational product
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study and/or poses difficulties in the interpretation of eventual changes occurring during the study
* Have systolic blood pressure of >140 millimeters of mercury (mmHg) or diastolic blood pressure of >90 mmHg
* Have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Show evidence of human immunodeficiency virus infection (HIV) and/or positive human HIV antibodies
* Show evidence of hepatitis C and/or positive hepatitis C antibody
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen
* Are women with a positive pregnancy test or women who are lactating
* Have used or intend to use over-the-counter or prescription medication within 14 days prior to dosing unless deemed acceptable by the investigator and sponsor's medical monitor
* Use of any drugs or substances that are known to be an inducer or inhibitor of cytochrome p450 3A4 (CYP3A4) (for example, St. John's wort) within 30 days prior to first dose of study drug
* Have donated blood of more than 500 milliliters (mL) within 30 days prior to first dose of study drug
* Have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females) or are unwilling to stop alcohol consumption for the duration of the study (1 unit equals 12 ounces [oz] or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits)
* Consume 5 or more cups of coffee (or other beverages of comparable caffeine content) per day, on a habitual basis, or any subjects unwilling to adhere to study caffeine restriction
* Have a daily use of greater than or equal to 5 tobacco- or nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) and are unwilling to refrain from using any tobacco- or nicotine-containing products within 7 days prior to first dose through the follow-up visit
* Have consumed grapefruit, grapefruit juice, Seville orange, Seville orange juice, or starfruit or products that contain these fruits within 7 days prior to first dose and during the study
* Unwilling to refrain from daily consumption of black licorice containing glycyrrhizic acid (that is, real licorice)
* In the opinion of the investigator or sponsor, are unsuitable for inclusion in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2011-10; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri, 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daytona Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a 2-part study, multiple ascending dose (MAD) and drug drug interaction (DDI). Participants were randomized to (Part 1) to 4 cohorts (Cohorts A through D) and randomized to receive either LY2484595 (5 ascending dose levels) or placebo. Cohort A consisted of 2 periods separated by a washout period of 14 days. DDI had 2 periods.
Groups:
- Part 1 Cohort A Sequence 1: Period 1:
  LY2484595: 100 milligrams (mg), tablets, oral administration, once daily (QD) on Days 1 through 14 of Period 1.
  Washout period lasting ≥14 days.
  Period 2:
  LY2484595: 1800 mg, tablets, oral administration, QD on Days 1 through 14 of Period 2.
- Part 1 Cohort A Sequence 2: Period 1:
  Placebo: dose-matched tablets, oral administration, once daily (QD) on Days 1 through 14 of Period 1.
  Washout period lasting ≥ 14 days
  Period 2:
  LY2484595: 1800 mg, tablets, oral administration, QD on Days 1 through 14 of Period 2.
- Part 1 Cohort A Sequence 3: Period 1:
  LY2484595: 100 milligrams (mg), tablets, oral administration, once daily (QD) on Days 1 through 14 of Period 1
  Washout period lasting ≥14 days
  Period 2:
  Placebo: tablets, oral administration, QD on Days 1 through 14 of Period 2
- Part 1 (Cohorts B Through D): Placebo: Placebo: tablets, oral administration, once daily (QD) on Days 1 through 14.
- Part 1 Cohort B: LY2484595: 300 milligrams (mg), tablets, oral administration, once daily (QD) on Days 1 through 14.
- Part 1 Cohort C: LY2484595: 600 milligrams (mg), tablets, oral administration, once daily (QD) on Days 1 through 14.
- Part 1 Cohort D: LY2484595: 1200 milligrams (mg), tablets, oral administration, once daily (QD) on Days 1 through 14.
- Part 2 Cohort E: Period 1:
  LY2484595: 100 milligrams (mg), tablet, oral administration, single dose on Day 1 of Period 1.
  Washout period lasting ≥ 14 days
  Period 2:
  Ketoconazole: 400 mg, tablet, oral administration, once daily (QD) on Days 1 through 14 of Period 2.
  LY2484595: 100 mg, tablet, oral administration, single dose on Day 5 of Period 2.
Period: Part 1 Period 1: Multiple Ascending Dose
Arm/Group | Part 1 Cohort A Sequence 1 | Part 1 Cohort A Sequence 2 | Part 1 Cohort A Sequence 3 | Part 1 (Cohorts B Through D): Placebo | Part 1 Cohort B | Part 1 Cohort C | Part 1 Cohort D | Part 2 Cohort E
Started | 12 | 4 | 4 | 10 | 16 | 12 | 12 | 0
Received at Least 1 Dose of Study Drug | 12 | 4 | 4 | 10 | 16 | 12 | 12 | 0
Completed | 12 | 4 | 4 | 9 | 14 | 10 | 11 | 0
Not Completed | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Part 1: Washout Period
Arm/Group | Part 1 Cohort A Sequence 1 | Part 1 Cohort A Sequence 2 | Part 1 Cohort A Sequence 3 | Part 1 (Cohorts B Through D): Placebo | Part 1 Cohort B | Part 1 Cohort C | Part 1 Cohort D | Part 2 Cohort E
Started | 12 | 4 | 4 | 0 (Participants in Part 1 Cohorts B through D participated in Period 1 only.) | 0 (Participants in Part 1 Cohort B participated in Period 1 only.) | 0 (Participants in Part 1 Cohort C participated in Period 1 only.) | 0 (Participants in Part 1 Cohort D participated in Period 1 only.) | 0
Completed | 11 | 4 | 4 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1 Period 2: Multiple Ascending Dose
Arm/Group | Part 1 Cohort A Sequence 1 | Part 1 Cohort A Sequence 2 | Part 1 Cohort A Sequence 3 | Part 1 (Cohorts B Through D): Placebo | Part 1 Cohort B | Part 1 Cohort C | Part 1 Cohort D | Part 2 Cohort E
Started | 11 | 4 | 4 | 0 (Participants in Part 1 Cohorts B through D participated in Period 1 only.) | 0 (Participants in Part 1 Cohort B participated in Period 1 only.) | 0 (Participants in Part 1 Cohort C participated in Period 1 only.) | 0 (Participants in Part 1 Cohort D participated in Period 1 only.) | 0
Received at Least 1 Dose | 11 | 4 | 4 | 0 | 0 | 0 | 0 | 0
Completed | 11 | 4 | 4 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 Period 1: Drug-drug Interaction
Arm/Group | Part 1 Cohort A Sequence 1 | Part 1 Cohort A Sequence 2 | Part 1 Cohort A Sequence 3 | Part 1 (Cohorts B Through D): Placebo | Part 1 Cohort B | Part 1 Cohort C | Part 1 Cohort D | Part 2 Cohort E
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12
Received at Least 1 Dose of Study Drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Part 2: Washout Period
Arm/Group | Part 1 Cohort A Sequence 1 | Part 1 Cohort A Sequence 2 | Part 1 Cohort A Sequence 3 | Part 1 (Cohorts B Through D): Placebo | Part 1 Cohort B | Part 1 Cohort C | Part 1 Cohort D | Part 2 Cohort E
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 Period 2: Drug-drug Interaction
Arm/Group | Part 1 Cohort A Sequence 1 | Part 1 Cohort A Sequence 2 | Part 1 Cohort A Sequence 3 | Part 1 (Cohorts B Through D): Placebo | Part 1 Cohort B | Part 1 Cohort C | Part 1 Cohort D | Part 2 Cohort E
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11
Received at Least 1 Dose of Study Drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11
Completed Dosing on Day 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- Part 1 (Cohort A) Sequence 1: Participants received 100 milligrams (mg) LY2484595 (tablets, oral administration) QD on Days 1 through 14. Then, received 1800 mg LY2484595 QD on Days 1 through 14 period 2.
- Part 1 (Cohort A) Sequence 2: Placebo: tablets, oral administration, once daily (QD) on Days 1 through 14 of Period 1 and 1800 mg LY2484595 on Days 1 through 14 of Period 2).
- Part 1 (Cohort A) Sequence 3: Participants received 100 mg LY2484595 (tablets, oral administration) once daily (QD) on Days 1 through 14. Then, received placebo QD on Days 1 through 14 period 2.
- Part 1 (Cohort B Through D) Placebo: Placebo: tablets, oral administration, once daily (QD) on Days 1 through 14.
- Part 1 (Cohort B): Participants received 300 mg LY2484595 (tablets, oral administration) QD on Days 1 through 14.
- Part 1 (Cohort C): Participants received 600 mg LY2484595 (tablets, oral administration) QD on Days 1 through 14.
- Part 1 (Cohort D): Participants received 1200 mg LY2484595 (tablets, oral administration) QD on Days 1 through 14.
- Part 2 (Cohort E): Participants received 100 mg LY2484595 (tablet, oral administration) as a single dose on Day 1 of Period 1. After a washout period lasting ≥14 days, participants received 400 mg ketoconazole (tablet, oral administration, QD) on Days 1 through 4 of Period 2, 400 mg ketoconazole (tablet, oral administration) and 100 mg LY2484595 (tablet, oral administration) on Day 5 of Period 2, and 400 mg ketoconazole (tablet, oral administration, QD) on Days 6 through 14 of Period 2.
- Total: Total of all reporting groups
Arm/Group | Part 1 (Cohort A) Sequence 1 | Part 1 (Cohort A) Sequence 2 | Part 1 (Cohort A) Sequence 3 | Part 1 (Cohort B Through D) Placebo | Part 1 (Cohort B) | Part 1 (Cohort C) | Part 1 (Cohort D) | Part 2 (Cohort E) | Total
Number analyzed (Participants) | 12 | 4 | 4 | 10 | 16 | 12 | 12 | 12 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (11.6) | 31.3 (3.9) | 41.8 (7.4) | 39.4 (13.7) | 41.1 (14.3) | 39.1 (10.7) | 45.8 (11.0) | 36.6 (7.9) | 39.8 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 0 | 3 | 5 | 2 | 2 | 3 | 19
  Male | 9 | 3 | 4 | 7 | 11 | 10 | 10 | 9 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 1 | 3 | 4 | 6 | 8 | 5 | 7 | 41
  Not Hispanic or Latino | 5 | 3 | 1 | 6 | 10 | 4 | 7 | 5 | 41
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 1 | 3 | 5 | 2 | 1 | 5 | 21
  White | 9 | 2 | 3 | 7 | 9 | 10 | 8 | 5 | 53
  More than one race | 0 | 1 | 0 | 0 | 2 | 0 | 3 | 0 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 4 | 4 | 10 | 16 | 12 | 12 | 12 | 82

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With 1 or More Adverse Events (AEs) or Any Serious AEs
Description: The number of participants with 1 or more AEs is summarized cumulatively. In addition, the number of participants with any serious AEs is summarized cumulatively. A serious AE is defined as an event that results in death, initial or prolonged hospitalization, is life-threatening, leads to persistent or significant disability/incapacity, is associated with congenital anomaly/birth defect, or is considered significant by the investigator for any other reason. A summary of serious and other non-serious AEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: Part 1: Baseline through ≥14 days after last dose of study drug (≥Day 28)
Population: All participants who received at least 1 dose of study drug.
Measure: Number; unit: Participants
Groups:
- Part 1 (Cohorts A Through D): Placebo: Placebo: tablets, oral administration, once daily (QD) on Days 1 through 14 of Period 1 (all cohorts) and Days 1 through 14 of Period 2 (Cohort A only)
- Part 1, Period 1 (Cohort A): 100 mg LY2484595: LY2484595: 100 milligrams (mg), tablets, oral administration, once daily (QD) on Days 1 through 14 of Period 1
- Part 1 (Cohort B): 300 mg LY2484595: LY2484595: 300 milligrams (mg), tablets, oral administration, once daily (QD) on Days 1 through 14
- Part 1 (Cohort C): 600 mg LY2484595: LY2484595: 600 milligrams (mg), tablets, oral administration, once daily (QD) on Days 1 through 14
- Part 1 (Cohort D): 1200 mg LY2484595: LY2484595: 1200 milligrams (mg), tablets, oral administration, once daily (QD) on Days 1 through 14
- Part 1, Period 2 (Cohort A): 1800 mg LY2484595: LY2484595: 1800 milligrams (mg), tablets, oral administration, once daily (QD) on Days 1 through 14 of Period 2
Arm/Group | Part 1 (Cohorts A Through D): Placebo | Part 1, Period 1 (Cohort A): 100 mg LY2484595 | Part 1 (Cohort B): 300 mg LY2484595 | Part 1 (Cohort C): 600 mg LY2484595 | Part 1 (Cohort D): 1200 mg LY2484595 | Part 1, Period 2 (Cohort A): 1800 mg LY2484595
Number analyzed (Participants) | 18 | 16 | 16 | 12 | 12 | 15
Participants
  AEs | 7 | 2 | 4 | 2 | 6 | 11
  Serious AEs | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Pharmacokinetics: Maximum Observed Plasma Concentration (Cmax) of LY2484595
Description: The geometric least squares (LS) means for the maximum observed plasma concentration (Cmax) of LY2484595 following administration of LY2484595 alone and with ketoconazole are reported. Least squares means were calculated from an analysis of variance (ANOVA) model with a fixed effect for treatment and a random effect for participant. The LS means for each treatment and the 90% confidence intervals (CI) for the difference in means were back transformed from the log scale to provide estimates of the geometric means and 90% CIs for the ratio of the geometric means (LY2484595 coadministered with ketoconazole and LY2484595 alone).
Time Frame: Part 2, Period 1, Day 1 through Day 8: Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168 Hours Post Dose; Period 2, Day 5 through Day 15: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240 Hours Post Dose
Population: Participants who received at least 1 dose of LY2484595 and had evaluable LY2484595 concentration data.
Measure: Least Squares Mean (90% Confidence Interval); unit: Nanograms per milliliter (ng/mL)
Groups:
- Part 2, Period 1: 100 mg LY2484595; Part 2, Period 2: 100 mg LY2484595 + 400 mg Ketoconazole: Period 1:
  LY2484595: 100 milligrams (mg), tablet, oral administration, single dose on Day 1 of Period 1
  Washout period lasting ≥ 14 days
  Period 2:
  Ketoconazole: 400 mg, tablet, oral administration, once daily (QD) on Days 1 through 14 of Period 2
  LY2484595: 100 mg, tablet, oral administration, single dose on Day 5 of Period 2
Arm/Group | Part 2, Period 1: 100 mg LY2484595 | Part 2, Period 2: 100 mg LY2484595 + 400 mg Ketoconazole
Number analyzed (Participants) | 12 | 10
Nanograms per milliliter (ng/mL) | 331.83 [236.06 to 466.45] | 643.99 [448.78 to 924.12]
Statistical Analysis 1: Comparison: Part 2, Period 1: 100 mg LY2484595 vs Part 2, Period 2: 100 mg LY2484595 + 400 mg Ketoconazole; Test type: Non-Inferiority or Equivalence — Up to 12 participants were enrolled in order for 8 to complete the study. The estimated variability in area under the concentration-time curve (AUC) was 20% coefficient of variation following a single dose of 100 mg LY2484595. Assuming that 70% of the total variability is contributed by intra-participant variability, a sample size of 8 participants provides a precision of ~15% for the geometric means ratio in AUC and Cmax of LY2484595 + ketoconazole to LY2484595 alone in log scale; Ratio of Geometric LS Means = 1.94, 90% CI 2-sided [1.39 to 2.72]

3. Primary Outcome: Pharmacokinetics: Time of Maximum Observed Plasma Concentration (Tmax) of LY2484595
Description: The median times to maximum observed plasma concentration (Tmax) of LY2484595 following administration of LY2484595 alone and with ketoconazole are reported.
Time Frame: as for outcome 2
Population: Participants who received at least 1 dose of LY2484595 and had evaluable LY2484595 concentration data.
Measure: Median (Full Range); unit: Hours (h)
Groups:
- Part 2, Period 1: 100 mg LY2484595; Part 2, Period 2: 100 mg LY2484595 + 400 mg Ketoconazole: Period 1:
  LY2484595: 100 milligrams (mg), tablet, oral administration, single dose on Day 1 of Period 1
  Washout period lasting ≥ 14 days
  Period 2:
  Ketoconazole: 400 mg, tablet, oral administration, once daily (QD) on Days 1 through 14 of Period 2.
  LY2484595: 100 mg, tablet, oral administration, single dose on Day 5 of Period 2
Arm/Group | Part 2, Period 1: 100 mg LY2484595 | Part 2, Period 2: 100 mg LY2484595 + 400 mg Ketoconazole
Number analyzed (Participants) | 10 | 10
Hours (h) | 3.00 [2.00 to 4.00] | 3.00 [2.00 to 3.00]
Statistical Analysis 1: Comparison: Part 2, Period 1: 100 mg LY2484595 vs Part 2, Period 2: 100 mg LY2484595 + 400 mg Ketoconazole; Test type: Superiority or Other; p = 1.0000, Wilcoxon signed rank; Median Difference (Final Values) = 0.00, 90% CI 2-sided [-0.50 to 0.50]

4. Primary Outcome: Pharmacokinetics: Area Under the Concentration-time Curve (AUC) of LY2484595
Description: The geometric least squares (LS) means of area under the concentration-time curve (AUC) from time zero extrapolated to infinity (AUC0-∞) of LY2484595 following administration of LY2484595 alone and with ketoconazole are reported. Least squares means were calculated from an analysis of variance (ANOVA) model with a fixed effect for treatment and a random effect for participant. The LS means for each treatment and the 90% confidence intervals (CI) for the difference in means were back transformed from the log scale to provide estimates of the geometric means and 90% CIs for the ratio of the geometric means (LY2484595 coadministered with ketoconazole and LY2484595 alone).
Time Frame: as for outcome 2
Population: Participants who received at least 1 dose of LY2484595 and had at least 3 consecutive plasma LY2484595 concentrations above the lower limit of quantification with at least 1 of these concentrations following the maximum observed plasma concentration (Cmax).
Measure: Geometric Mean (90% Confidence Interval); unit: Nanograms * hours per milliliter
Arm/Group | Part 2, Period 1: 100 mg LY2484595 | Part 2, Period 2: 100 mg LY2484595 + 400 mg Ketoconazole
Number analyzed (Participants) | 12 | 9
Nanograms * hours per milliliter | 5265 [4106 to 6751] | 12471 [9422 to 16508]
Statistical Analysis 1: Comparison: Part 2, Period 1: 100 mg LY2484595 vs Part 2, Period 2: 100 mg LY2484595 + 400 mg Ketoconazole; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Ratio of Geometric LS means = 2.37, 90% CI 2-sided [1.77 to 3.18]

5. Secondary Outcome: Pharmacodynamics: Change From Baseline to Day 21 in Cholesteryl Ester Transfer Protein (CETP) Activity
Time Frame: Day 1 (Baseline) and Day 21
Population: Participants who received at least 1 dose of LY2484595 or placebo and had evaluable pharmacodynamic (CETP) data.
Measure: Mean (Standard Deviation); unit: Picomoles per milliliters per minute
Arm/Group | Part 1 (Cohorts A Through D): Placebo | Part 1, Period 1 (Cohort A): 100 mg LY2484595 | Part 1 (Cohort B): 300 mg LY2484595 | Part 1 (Cohort C): 600 mg LY2484595 | Part 1 (Cohort D): 1200 mg LY2484595 | Part 1, Period 2 (Cohort A): 1800 mg LY2484595
Number analyzed (Participants) | 18 | 16 | 15 | 11 | 11 | 15
Picomoles per milliliters per minute | 1.3 (6.9) | -0.4 (3.1) | -0.4 (6.3) | -9.1 (8.8) | -9.5 (5.0) | -12.9 (7.5)

6. Secondary Outcome: Pharmacodynamics: Change From Baseline to Day 21 in High-density Lipoprotein Cholesterol (HDL-C), Low-density Lipoprotein Cholesterol (LDL-C), and Triglycerides (TG)
Time Frame: Day 1 (Baseline) and Day 21
Population: Participants who received at least 1 dose of LY2484595 or placebo during Period 1 and had evaluable pharmacodynamic (HDL-C, LDL-C, TG) data.
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Groups:
- Part 1, Period 1 (Cohorts A Through D): Placebo: Placebo: tablets, oral administration, once daily (QD) on Days 1 through 14 of Period 1 (all cohorts)
Arm/Group | Part 1, Period 1 (Cohorts A Through D): Placebo | Part 1, Period 1 (Cohort A): 100 mg LY2484595 | Part 1 (Cohort B): 300 mg LY2484595 | Part 1 (Cohort C): 600 mg LY2484595 | Part 1 (Cohort D): 1200 mg LY2484595
Number analyzed (Participants) | 14 | 16 | 15 | 11 | 11
Millimoles per liter (mmol/L)
  HDL-C | -0.08 (0.17) | 0.35 (0.22) | 0.49 (0.31) | 0.77 (0.49) | 0.80 (0.22)
  LDL-C | -0.42 (0.74) | -0.16 (0.31) | -0.48 (0.55) | -1.15 (0.93) | -1.01 (0.57)
  TG | 0.56 (0.87) | 0.55 (0.81) | 0.44 (0.61) | 0.26 (0.38) | 0.52 (0.57)

7. Secondary Outcome: Pharmacokinetics: Maximum Observed Plasma Concentration (Cmax) of LY2484595
Description: The maximum observed plasma concentrations (Cmax) of LY2484595 after a single dose and after once daily (QD) dosing for 14 consecutive days are reported.
Time Frame: Part 1, Periods 1 and 2, Day 1: Predose, 1, 2, 3, 4, 6, 8, 12, and 24 Hours Postdose; Day 14 through Day 21: Predose, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 168 Hours Post Dose
Population: Participants who received at least 1 dose of LY2484595 and had evaluable LY2484595 concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Part 1, Period 1 (Cohort A): 100 mg LY2484595 | Part 1 (Cohort B): 300 mg LY2484595 | Part 1 (Cohort C): 600 mg LY2484595 | Part 1 (Cohort D): 1200 mg LY2484595 | Part 1, Period 2 (Cohort A): 1800 mg LY2484595
Number analyzed (Participants) | 16 | 16 | 12 | 12 | 15
Nanograms per milliliter (ng/mL)
  Day 1 | 628 (79) | 1990 (60) | 2720 (59) | 4450 (53) | 3580 (73)
  Day 14: number analyzed (Participants) | 16 | 15 | 12 | 11 | 15
  Day 14 | 978 (41) | 1970 (37) | 4180 (42) | 5410 (48) | 5750 (35)

8. Secondary Outcome: Pharmacokinetics: Time of Maximum Observed Plasma Concentration (Tmax) of LY2484595
Description: The times of maximum observed plasma concentrations (tmax) of LY2484595 after a single dose and after once daily (QD) dosing for 14 consecutive days are reported.
Time Frame: as for outcome 7
Population: Participants who received at least 1 dose of study drug and had evaluable LY2484595 concentration data.
Measure: Median (Full Range); unit: Hours (h)
Arm/Group | Part 1, Period 1 (Cohort A): 100 mg LY2484595 | Part 1 (Cohort B): 300 mg LY2484595 | Part 1 (Cohort C): 600 mg LY2484595 | Part 1 (Cohort D): 1200 mg LY2484595 | Part 1, Period 2 (Cohort A): 1800 mg LY2484595
Number analyzed (Participants) | 16 | 16 | 12 | 12 | 15
Hours (h)
  Day 1 | 3.00 [2.00 to 8.00] | 3.00 [1.00 to 8.00] | 3.00 [2.00 to 4.00] | 2.00 [1.00 to 8.00] | 2.00 [1.00 to 4.00]
  Day 14: number analyzed (Participants) | 16 | 15 | 12 | 11 | 15
  Day 14 | 4.00 [2.00 to 6.00] | 2.00 [2.00 to 4.00] | 2.50 [1.00 to 4.00] | 2.00 [1.00 to 6.00] | 3.00 [1.00 to 6.00]

9. Secondary Outcome: Pharmacokinetics: Area Under the Concentration-time Curve (AUC) of LY2484595
Description: Exposure to LY2484595 in terms of the area under the concentration-time curves (AUC) after a single dose and after once daily (QD) dosing for 14 consecutive days are reported.
Time Frame: as for outcome 7
Population: All participants who received at least 1 dose of LY2484595 and had at least 3 consecutive plasma LY2484595 concentrations above the lower limit of quantification with at least 1 of these concentrations following the maximum observed plasma concentration (Cmax).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms * hour per milliliter
Groups:
- Part 1, Period 2 (Cohort A): 1800 mg LY2484595: LY284595: 1800 milligrams (mg), tablets, oral administration, once daily (QD) on Days 1 through 14 of Period 2
Arm/Group | Part 1, Period 1 (Cohort A): 100 mg LY2484595 | Part 1 (Cohort B): 300 mg LY2484595 | Part 1 (Cohort C): 600 mg LY2484595 | Part 1 (Cohort D): 1200 mg LY2484595 | Part 1, Period 2 (Cohort A): 1800 mg LY2484595
Number analyzed (Participants) | 16 | 16 | 12 | 12 | 15
Nanograms * hour per milliliter
  Day 1 | 4780 (57) | 14500 (47) | 21300 (55) | 36300 (46) | 31300 (63)
  Day 14: number analyzed (Participants) | 16 | 15 | 12 | 11 | 15
  Day 14 | 8110 (30) | 17900 (27) | 36200 (38) | 46900 (43) | 56600 (30)

ADVERSE EVENTS:
Description: All randomized participants who received at least 1 dose of study drug.
Groups:
- Part 1 (Cohorts A Through D): Placebo: tablets, oral administration, once daily (QD) on Days 1 through 14 of Period 1 (all cohorts) and Days 1 through 14 of Period 2 (Cohort A only)
- Part 1, Period 1 (Cohort A): LY2484595: 100 milligrams (mg), tablets, oral administration, once daily (QD) on Days 1 through 14 of Period 1
- Part 1, Period 2 (Cohort A): LY284595: 1800 milligrams (mg), tablets, oral administration, once daily (QD) on Days 1 through 14 of Period 2
- Part 2, Period 2: 400 mg Ketoconazole; Part 2, Period 2: 100 mg LY2484595 + 400 mg Ketoconazole: Period 1:
  LY2484595: 100 milligrams (mg), tablet, oral administration, single dose on Day 1 of Period 1
  Washout period lasting ≥ 14 days
  Period 2:
  Ketoconazole: 400 mg, tablet, oral administration, once daily (QD) on Days 1 through 14 of Period 2
  LY2484595: 100 mg, tablet, oral administration, single dose on Day 5 of Period 2
Arm/Group | Part 1 (Cohorts A Through D) | Part 1, Period 1 (Cohort A) | Part 1, Period 2 (Cohort A) | Part 1 (Cohort B): 300 mg LY2484595 | Part 1 (Cohort C): 600 mg LY2484595 | Part 1 (Cohort D): 1200 mg LY2484595 | Part 2, Period 1: 100 mg LY2484595 | Part 2, Period 2: 400 mg Ketoconazole | Part 2, Period 2: 100 mg LY2484595 + 400 mg Ketoconazole
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/16 | 0/15 | 0/16 | 0/12 | 0/12 | 0/12 | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 7/18 | 2/16 | 11/15 | 4/16 | 2/12 | 6/12 | 4/12 | 5/11 | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 (Cohorts A Through D) (N=18) | Part 1, Period 1 (Cohort A) (N=16) | Part 1, Period 2 (Cohort A) (N=15) | Part 1 (Cohort B): 300 mg LY2484595 (N=16) | Part 1 (Cohort C): 600 mg LY2484595 (N=12) | Part 1 (Cohort D): 1200 mg LY2484595 (N=12) | Part 2, Period 1: 100 mg LY2484595 (N=12) | Part 2, Period 2: 400 mg Ketoconazole (N=11) | Part 2, Period 2: 100 mg LY2484595 + 400 mg Ketoconazole (N=10)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 6 (7) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 10 (13) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 6 (9) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Oedema mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral mucosal erythema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling jittery (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritability (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 6 (16) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 4 (5) | 0 (0)
Muscle contractions involuntary (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Capillary fragility (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less